CLINICAL TRIAL: NCT06109324
Title: A Multicenter Randomized Controlled Trial on the Effects of Upper Limb Robotic Rehabilitation on Sensory and Cognitive Impairments in Subjects With Stroke. The SCORES (Sensory and Cognitive Outcomes of Robotic Exercises in Stroke) Study.
Brief Title: Sensory and Cognitive Outcomes of Robotic Exercises in Stroke (SCORES)
Acronym: SCORES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: IRCCS Centro Neurolesi Bonino Pulejo (Other); Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCORES_clinicalstudy
Record Dates: First submitted 2023-10-23; First posted 2023-10-31 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: robotics; cognition; rehabilitation; upper extremity; sensorimotor
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic Rehabilitation (Experimental)
  Interventions: Other: Robotic Rehabilitation of the upper limb
- Conventional treatment (Active Comparator)
  Interventions: Other: Conventional Rehabilitation of the upper limb

INTERVENTIONS:
Other: Robotic Rehabilitation of the upper limb — Upper limb rehabilitation using a set of 4 devices. A set of motor/cognitive exercises will be selected to train also attention, memory, executive function, speed of processing, and visuospatial abilities.The following devices will be used: (a) a robotic device that allows passive, active, and active-assistive planar movements of the shoulder and elbow joints (Motore, Humanware); (b) a robotic device that allows passive, active, and active-assistive finger flexion and extension movements (Amadeo, Tyromotion); (c) a sensor-based system that allows unsupported 3-dimensional movements of shoulder, elbow, and wrist joint, both unimanual and bimanual (Pablo, Tyromotion); and (d) a robotic system that allows 3-dimensional, unimanual and bimanual, movements of the shoulder joint, with arm weight support (Diego, Tyromotion).
  The rehabilitation treatment will be performed daily for 45 minutes, 5 days/week, for a total of 30 sessions.
  Arms: Robotic Rehabilitation
Other: Conventional Rehabilitation of the upper limb — Upper limb rehabilitation using conventional techniques, focused on upper limb reprogramming sensorimotor function, hypertonus, inhibition and functional improvement.
  The rehabilitation treatment will be performed daily for 45 minutes, 5 days/week, for a total of 30 sessions.
  Arms: Conventional treatment

SUMMARY:
Based on the findings of meta-analyses, upper limb robotic rehabilitation has shown to enhance daily living activities, motor function, and strength in stroke patients. However, when compared to traditional methods, recent randomized controlled trials conducted on larger participant groups failed to identify significant differences in motor-related outcomes between the two approaches.

In addition to motor deficits, stroke survivors often experience cognitive decline and sensory disturbances, which can significantly impede their recovery process. The introduction of multisensory stimulation and an enriched environment through robotic interventions may offer valuable supplementary treatments in these specific areas. Nevertheless, this aspect of treatment has not been thoroughly explored.

This study seeks to assess the effectiveness of upper limb robotic rehabilitation in individuals recovering from subacute strokes, in comparison to conventional treatments. Specifically, it aims to determine whether this robotic therapy can lead to improvements in (a) cognitive deficits, (b) somatosensory impairment, and (c) how these sensory and cognitive deficits influence the process of motor recovery.

DETAILED DESCRIPTION:
The study aims to investigate whether an upper limb robotic treatment could have a greater impact than a conventional approach on specific cognitive domains in patients with stroke, as well as in restoring the somatosensory impairment in patients with stroke.

For this aim, 126 consecutive subjects with stroke in the sub-acute phase (within 6 months after stroke) will be enrolled and randomized to either the robotic (RG) or the conventional group (CG). The sample size was calculated by means of a 2- sided, 2-sample t-test assuming: 80% power; type I error of 0.05; a mean difference of 2.15 units on the MoCA, a common standard deviation of 3.77 points (Wu 2019). Considering a dropout rate of 20%, the final sample size required was estimated to be 126 subjects.

Randomization will be stratified according to a cut-off of 18.28 on the MoCA demographically adjusted total score (inner confidence limit of the 5th centile of the normal population) indicating a borderline performance, to ensure that the subjects' characteristics in each group will be closely matched. In the RG, patients will undergo robotic therapy, while a conventional approach will be used in the CG. The rehabilitation treatments, either robotic or conventional, will be performed daily for 45 minutes, 5 days/week, for a total of 30 sessions. Patients in the RG will be treated using a set of devices that allow bi- and three-dimensional movements of the shoulder, elbow, wrist, and fingers (Aprile et al, 2019). Motor and cognitive tasks, carefully selected among those available, will be performed during the treatment, following a protocol already proposed in a previous pilot study (Aprile et al, 2021). Visual and auditory feedback will be provided to help the patients. In the RG, treatment will focus on reprogramming sensorimotor function, hypertonus inhibition, and functional improvement. Patients will be evaluated at baseline (T0), the end of the rehabilitation protocol (T1), and a 6-month follow-up (T2).

ELIGIBILITY:
Inclusion Criteria:

* a single event, verified by MRI or CT;
* age between 18 and 85 years;
* time since stroke within six months;
* a demographically adjusted total score of the Montreal Cognitive Assessment (MoCA) between 15.5 and 22.23

Exclusion Criteria:

* behavioural and cognitive disorders and/or reduced compliance that would interfere with active therapy;
* fixed contraction deformity in the affected limb that would interfere with active therapy (ankylosis, Modified Ashworth Scale = 4);
* severe deficits in visual acuity.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Montreal Cognitive Assessment | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention
  It is a validated test of cognitive impairment. It ranges from 0 (indicating worse cognitive function) to 30 (best cognitive function).

SECONDARY OUTCOMES:
Changes in Montreal Cognitive Assessment | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  It is a validated test of cognitive impairment. It ranges from 0 (indicating worse cognitive function) to 30 (best cognitive function).
Changes in Symbol Digit Modalities Test | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The Symbol Digit Modalities Test evaluates information processing speed. It consists of a simple task of replacing symbols with numbers. Using a reference key, the patient has 90 seconds to match a sequence of symbols with the correspondent numbers as rapidly as possible. Both written or oral administration can be used.
  For each correct answer, a point is assigned.
Changes in Tower of London | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The Tower of London test is a tool to assess strategic decision and problem solving. The patient is required to move different colored balls on the three pegs of different lengths, according to a model and a number of established moves. The maximum time for each configuration is 60 seconds.
Changes in Rey-Osterrieth Complex Figure test | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The Rey-Osterrieth Complex Figure is a neuropsychological assessment for evaluation of visuospatial abilities, memory, attention, planning, working memory and executive functions. The patient is required to copy a complex figure freehand (recognition), and then draw it from memory (recall). The score is assigned based on the correctness of each line (from 0 to 2)
Changes in Visual search test | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  It is a validated measure of visual attention.
Changes in Fugl-Meyer Assessment of the Upper Extremity (motor score) | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  It is a stroke-specific, performance-based impairment index. It ranges from 0 (hemiplegia) to 66 points (normal).
Changes in Thumb Localizing Test | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  It is a standardised measure of proprioception. It ranges from 0 (normal) to 3.
Changes in Semmes Weinstein filament test | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  It measure the level of light touch sensation of the tips of the thumb and index finger. The Semmes Weinstein filament test kit consists of 20 flexible nylon monofilaments of constant length, but varying in diameter. They are labeled so as to give a linear scale of perceived intensity (1.65-6.65) using a logarithmic scale of applied force: labeled number = Log10 of (10 × force in milligrams). The more the labeled number increases, the thicker the filament becomes, and the more pressure is necessary to bend the filament.
Changes in Fugl-Meyer Assessment of the Upper Extremity (sensation score) | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  It is a stroke-specific, performance-based impairment index. It ranges from 0 (no sensation) to 12 points (normal).
Changes in Box and Block test | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The Box and Block test is a standard measure for evaluating manual dexterity. The participants grasp and transfer one-inch square blocks from one compartment to the other, transferring as many as possible. The number of blocks transferred from one side to the other within 1 min is recorded.
Changes in Motricity Index | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  It is a validated measure of upper limb strength. It ranges from 0 (worse) to 100 (normal strength).
Changes in Modified Barthel Index | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The modified is an ordinal scale used to measure performance in activities of daily living. It ranges from 0 to 100, with lower scores indicating increased disability.
Changes in Numerical Rating Scale for Pain | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale, from 0 (no pain) to 10 (worst pain imaginable).
Changes in Neuropathic Pain Symptom Inventory | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  It is a validated scale for evaluating both peripheral and central neuropathic pain. It ranges from 0 to 100 (most imaginable pain)
Changes in Douleur Neuropathique 4 | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  It is a validated clinician-administered screening tool for neuropathic pain. It ranges from 0 to 10; higher values means higher neuropathic pain probability.
Changes in Post-stroke Depression Rating Scale | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  It is a validated measure of depression in post-stroke patients. The score ranges from 0 (best) to 45 (worse)
Changes in Intrinsic Motivation Inventory | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The Intrinsic Motivation Inventory (IMI) is a multidimensional measurement method designed to assess participants' subjective experience related to a target activity in laboratory experiments

OTHER OUTCOMES:
Changes in robotic score duration | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "Duration" is the time required to complete the task. It is measured in seconds
Changes in robotic score speed | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "Velocity_mean" is the average velocity of the device during the test. It is measured in m/s.
Changes in robotic score length | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "Length_tot" is the global length of the path travelled by the subject during center-out movements. It is measured in meters and it ranges from 0 (no movement) to 2.808 m (patient can fully perform the entire task).
Changes in robotic score useful work | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "useful work" is the amount of total work directed towards the target. It is measured in Joules.
Changes in robotic score strength | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The kinetics of the end-effector of the robot will be measured by the robot during reaching tasks performed by the patient against the device. The outcome will be the maximum values towards 8 targets
Changes in robotic score finger strength (flexion and extension) | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  It is the isometric strength for the hand, in both flexion and extension
Changes in robotic score muscle tone at rest | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  It is the passive baseline force of the finger muscles.
Changes in matching test mean error | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The mean value of the absolute differences between the actual and the desired positions.
Changes in matching test variability | Baseline, up to 7 days after the enrollment; up to 3 days after the intervention; 6 months after the end of the intervention
  The standard deviation of the matching errors across trials.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Germanotta, PhD, Study Director — IRCCS Fondazione Don Carlo Gnocchi
Locations (3):
- Italy (3):
  - IRCCS Fondazione Don Carlo Gnocchi, Florence
  - IRCCS Centro Neurolesi Bonino Pulejo, Messina
  - Fondazione Don Carlo Gnocchi - Centro Santa Maria della Provvidenza, Roma